CLINICAL TRIAL: NCT02000570
Title: Abilities of Dynamic Preload Dependence Indicators to Predict Fluid Responsiveness During Neurosurgery in Sitting Position
Brief Title: Dynamic Preload Indicators in Sitting Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013.813; 2013-A00937-38 (Other: ID-RCB)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Neurosurgery in Sitting Position
Keywords: sitting position; PPV; SVV; PVI; fluid challenge; preload indicators
MeSH Terms: interventions — Sitting Position; Neurosurgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sitting position (Experimental)
  Interventions: Procedure: Sitting position (neurosurgery)

INTERVENTIONS:
Procedure: Sitting position (neurosurgery)

SUMMARY:
Intraoperative optimization of cardiac output using goal directed fluid challenge is associated with better outcome. Dynamic preload dependence indicators are well validated during surgery in supine position. Positioning from supine to sitting position under anesthesia is responsible of several hemodynamic changes. Predictability and cut-off values of dynamic preload dependence indicators during surgery in sitting position are unknown. The objective of this prospective study is to evaluate ability of three dynamic preload dependence indicators, i.e. PPV (Pulse Pressure Variation), SVV (Stroke Volume Variation) and PVI (Plethysmographic Variability Index), during neurosurgery in sitting position.

DETAILED DESCRIPTION:
The primary objective is to determine PPV, SVV and PVI thresholds for which patients respond to fluid challenge in sitting position.

The secondary objectives are to determine variations of PPV, SVV and PVI measures before and after positioning in sitting position, and to compare these values to each other.

ELIGIBILITY:
Inclusion Criteria:

* neurosurgery in sitting position
* age > 18

Exclusion Criteria:

* arrhythmias
* severe heart failure
* severe lung disease
* contraindications to esophageal Doppler monitoring probe insertion (i.e. esophageal weakness)
* renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
PPV (Pulse pressure variation) | 3 minutes before and after fluid challenge in sitting position
  PPV is derived from arterial pressure waveforms and is displayed in real -time on Intellivue MP70 Philips monitors.
  Value will be recorded before fluid challenge. Responders will be assessed by esophageal Doppler.
SVV (Stroke volume variation) | 3 minutes before and after positioning in sitting position
  SVV is derived from arterial pressure waveforms and is displayed in real -time on Vigileo Edwards Lifesciences monitors.
  Value will be recorded before fluid challenge. Responders will be assessed by esophageal Doppler.
PVI (Plethysmographic variability index) | 3 minutes before and after positioning in sitting position
  PVI is derived from plethysmography waveforms and is displayed in real-time on Radical 7 Masimo monitors.
  Value of each indicator will be recorded before fluid challenge. Responders will be assessed by esophageal Doppler.

CONTACTS AND LOCATIONS:
Locations (1):
- Fédération d'anesthésie réanimation Hôpital Pierre Wertheimer, Bron, France